CLINICAL TRIAL: NCT01726712
Title: Network Supported Engagement In HIV Care
Acronym: NSEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); ACCESS Community Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-0654; 1R34MH097622-01 (NIH)
Record Dates: First submitted 2012-10-15; First posted 2012-11-15 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: HIV; Patient Acceptance of Health Care
Keywords: Patient Care Management; Primary Health Care; HIV; Patient Acceptance of Health Care
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine Care (No Intervention)
- Supportive Contact (Active Comparator)
  Interventions: Other: Supportive Care

INTERVENTIONS:
Other: Supportive Care — Provide emotional support. Provide practical support. Support friend/family by helping him find information or help for those with HIV in the community
  Arms: Supportive Contact

SUMMARY:
The Network Supported Engagement in Care (NSEC) intervention is a brief, theory based and culturally sensitive intervention designed to capitalize on organic yet underutilized social support networks in the lives of young black men who have sex with men (YBMSM) who have been recently diagnosed with HIV. The intervention has been developed with input from clients and their support network members, case managers, social workers, HIV primary care providers and pastoral care at a Federally Qualified Health Center. The goal of the intervention is to improve retention in care for newly diagnosed YBMSM who present for their first HIV primary care clinic appointment.

ELIGIBILITY:
Inclusion Criteria:

Index subjects

* Self-identify as African-American and male;
* same gender anal/oral sex in the past 2 years;
* English speaking;
* have at least one SC in their network;
* own a cell phone not shared with other persons;
* agreeable to text-message mini-booster sessions; and
* between the ages of 16-29 years old.

Supportive Contact:

* Index participant has agreed to including the supportive contact;
* Supportive contact is willing to attend face to face and telephone mini-booster sessions;
* 18 years of age or older;
* English speaking; and
* owns a cell phone that is not shared with other persons.

Exclusion Criteria:

Index Subject:

* unable to provide assent/consent;
* plan to move out of the area within the next 12 months;
* are not willing to attend intervention sessions; or
* not willing to return for assessments

Supportive Contact:

* unable to provide informed consent; or
* not willing to return for 3 and 12 month assessments.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Missed Visit Proportion (MVP) | 12 months
  The primary aim is to test for differences in MVP by treatment group across the study time period of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John A Schneider, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States